CLINICAL TRIAL: NCT00557310
Title: The Effects of Teriparatide on Bone Microarchitecture as Determined by High Resolution Magnetic Resonance Imaging and Digital Topological Analysis
Brief Title: A Study Using Imaging Technology to Measure Changes in Bone Structure After Treatment With Teriparatide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11996; B3D-US-GHDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-10

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: osteoporosis, teriparatide, postmenopausal, MRI, finite element analysis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teriparatide (Experimental): 20 micrograms (mcg) teriparatide subcutaneous injection per day for 18 months, with possibility to continue for 24 months
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — 20 mcg teriparatide subcutaneous injection per day for 18 months, with possibility to continue for 24 months
  Other Names: LY333334; FORTEO; FORSTEO

SUMMARY:
The purpose of this study is to use imaging technologies to demonstrate the effects of teriparatide on bone structure following 18 to 24 months of therapy in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
As teriparatide is approved for up to 24 months of treatment in the US, patients will be given the option to continue in a 6-month extension phase upon completion of 18 months of teriparatide treatment. This extension will allow for collection of additional bone quality data. In Canada, the use of teriparatide is currently approved for 18 months. Patients in Canada may be given the opportunity to participate in the 6-month extension phase, contingent upon Health Canada approval of the use of teriparatide treatment for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal (after the "change of life") women with osteoporosis
* between the ages of 45-85
* have low bone mass as determined by a bone density test
* have at least one prior atraumatic vertebral or nonvertebral fracture(with a T-score of -2.0 or lower at the lumbar spine, total hip, or femoral neck) or, no prior fracture (with a T-score of -3.0 or lower at these same sites)
* could have taken up to 5 years total of certain oral osteoporosis medications such as alendronate, risedronate, or ibandronate

Exclusion Criteria:

* have conditions that would affect the bone in the region of the wrist or have had a previous fracture of either wrist which might affect results of study
* have a metal implant or have had a hip replacement in either hip which might affect results of study
* have an increased risk of osteosarcoma; includes Paget's disease of bone, a previous bone tumor, or x-ray treatment to the skeleton
* currently have active or suspected diseases that affect the bone, other than osteoporosis
* have abnormal levels of calcium, parathyroid hormone in blood, or other laboratory values

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia, Canada

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the 18 month main study had an option to continue treatment for an additional 6 months (Extension Phase).
Groups:
- Teriparatide: 20 microgram (mcg) teriparatide subcutaneous injection per day for 18 months, with possibility to continue for 24 months
Period: Main Study (0 - 18 Months)
Arm/Group | Teriparatide
Started | 35
Completed | 30 (One had a metal hip implant, a protocol violation, and was excluded from efficacy analyses.)
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Period: Extension Phase (18 - 24 Months)
Arm/Group | Teriparatide
Started | 30
Completed | 25 (One had a metal hip implant, a protocol violation, and was excluded from efficacy analyses.)
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Teriparatide
Number analyzed (Participants) | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 61.96 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31
  Hispanic | 2
  West Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
  Canada | 6
Dominant Hand [Number; unit: participants]
  Left | 1
  Right | 33
Prevalent Fractures [Number; unit: participants] — A prevalent fracture is defined as a fracture that a participant already had at the time of study entry. One participant had both a vertebral and non-vertebral fracture and therefore the total number of participants is higher than the baseline population number.
  participants
    None | 14
    Any vertebral fracture | 4
    Any non-vertebral fracture | 17
Years Postmenopausal [Mean (Standard Deviation); unit: years] | 16.97 (12.10)
Prior Bisphosphonate Use [Number; unit: participants]
  Yes | 21
  No | 13
Lumbar Spine T-Score [Mean (Standard Deviation); unit: units on a scale] — The T-score is a comparison of a patient's bone mineral density (BMD) to that of the mean BMD for a healthy population of women at peak bone mass (30 years). A normal T-score has a value of -1.0 or higher. Osteoporosis is defined as a T-score of -2.5 or lower, meaning a bone mineral density that is two and a half standard deviations below the mean BMD of a healthy population of women at peak bone mass (30 years).
  units on a scale | -2.91 (1.04)
Femoral Neck T-Score [Mean (Standard Deviation); unit: units on a scale] | -2.38 (0.67)
Total Hip T-Score [Mean (Standard Deviation); unit: units on a scale] | -1.80 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Surface-to-Curve Ratio (SCR) in the Distal Radius at Month 18 Endpoint
Description: SCR is a measure of the computed ratio of plate-like to rod-like structures in a given volume of trabecular bone and reflects the integrity of the trabecular network. The higher the value for SCR, the more intact the trabecular network. Least squares (LS) mean of the percent change from baseline to 18 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 18 months
Population: Participants who were assigned to treatment, had non-missing baseline and at least one non-missing post-baseline measurement value.
Measure: Least Squares Mean (Standard Error); unit: percent (%) change of ratio
Arm/Group | Teriparatide
Number analyzed (Participants) | 25
percent (%) change of ratio | 4.53 (4.89)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.363, Mixed Model Repeated Measurements

2. Secondary Outcome: Percent Change From Baseline in Surface-to-Curve Ratio (SCR) in the Distal Radius at Month 24 Endpoint
Description: SCR is a measure of the computed ratio of plate-like to rod-like structures in a given volume of trabecular bone and reflects the integrity of the trabecular network. The higher the value for SCR, the more intact the trabecular network. Least squares (LS) mean of the percent change from baseline to 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of ratio
Arm/Group | Teriparatide
Number analyzed (Participants) | 21
% change of ratio | 1.44 (6.88)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.837, Mixed Model Repeated Measurements

3. Secondary Outcome: Percent Change From Baseline in Cortical Thickness (CT) in the Distal Radius at Month 18 and 24 Endpoint
Description: Cortical thickness (CT) is the thickness of both cortices in a given volume of bone. Least squares (LS) mean of the percent change from baseline to 18, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of millimeter (mm)
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of millimeter (mm)
  18 month percent change (n=25) | -0.61 (2.56)
  24 month percent change (n=21) | -0.22 (2.59)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.816, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.934, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 24 months

4. Secondary Outcome: Percent Change From Baseline in Topological Erosion Index (TEI) in the Distal Radius at Month 18 and 24 Endpoint
Description: TEI is the ratio of the sum of topological parameters expected to increase with bone erosion compared to the sum of those expected to decrease. The lower the value for TEI, the more intact the trabecular network. Least squares (LS) mean of the percent change from baseline to 18, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of ratio
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of ratio
  18 month percent change (n=25) | 3.36 (3.31)
  24 month percent change (n=21) | 8.46 (4.63)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.324, Mixed Model Repeated Measures — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.089, Mixed Model Repeated Measures — P-value is for the percent change from baseline at 24 months

5. Secondary Outcome: Percent Change From Baseline in Bone Volume (BV)/Total Volume (TV) Ratio in the Distal Radius at Month 18 and 24 Endpoint
Description: BV/TV is the estimate of the ratio of detectable bone relative to the total volume of the region of interest. Least squares (LS) mean of the percent change from baseline to 18, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of ratio
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of ratio
  18 month percent change (n=25) | 0.36 (1.85)
  24 month percent change (n=21) | -3.14 (2.40)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.847, Mixed Model Repeated Measurements; P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.212, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 24 months

6. Secondary Outcome: Percent Change From Baseline in Surface-to-Curve Ratio (SCR) at Month 3, 6, 12, 18 and 24 Endpoint
Description: SCR is a measure of the computed ratio of plate-like to rod-like structures in a given volume of trabecular bone and reflects the integrity of the trabecular network. The higher the value for SCR, the more intact the trabecular network. Least squares (LS) mean of the percent change from baseline to 3, 6, 12, 18, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 3, 6, 12, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of ratio
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of ratio
  3 month percent change (n=32) | -3.38 (3.46)
  6 month percent change (n=30) | 0.43 (4.05)
  12 month percent change (n=28) | 2.36 (4.56)
  18 month percent change (n=25) | 4.53 (4.89)
  24 month percent change (n=21) | 1.44 (6.88)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.335, Mixed Model Repeated Measurements; P-value is for the percent change from baseline at 3 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.916, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 6 months
Statistical Analysis 3: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.610, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 12 months
Statistical Analysis 4: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.363, Mixed Model Repeated Measurements; P-value is for the percent change from baseline at 18 months
Statistical Analysis 5: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.837, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 24 months

7. Secondary Outcome: Percent Change From Baseline in Volumetric Bone Mineral Density (BMD) of Lumbar Spine at Month 18 Endpoint
Description: Volumetric BMD is a measure of the amount of mineral in a given volume of bone, expressed as milligram per cubic centimeter (mg/cm³). Least squares (LS) mean of the percent change from baseline to 18 months is from an analysis of variance (ANOVA). The model included terms for investigator site and prior bisphosphonate use.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of mg/cm³
Arm/Group | Teriparatide
Number analyzed (Participants) | 28
% change of mg/cm³ | 10.05 (1.55)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, ANOVA

8. Secondary Outcome: Percent Change From Baseline in Volumetric Bone Mineral Density (BMD) of Hip at Month 18 Endpoint
Description: Volumetric BMD is a measure of the amount of mineral in a given volume of bone. Least squares (LS) mean of the percent change from baseline to 18 months is from an analysis of variance (ANOVA). The model included terms for investigator site and prior bisphosphonate use.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of mg/cm³
Arm/Group | Teriparatide
Number analyzed (Participants) | 25
% change of mg/cm³ | 2.22 (0.88)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.021, ANOVA

9. Secondary Outcome: Percent Change From Baseline in the Estimate of Bone Strength of Lumbar Spine at Month 18 Endpoint
Description: Finite Element Analysis of computed tomography (CT) data from spine is used to estimate the strength of a vertebral body using a virtual axial load. Least squares (LS) mean of the percent change from baseline to 18 months is from an analysis of variance (ANOVA). The model included terms for investigator site and prior bisphosphonate use.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of Newtons
Arm/Group | Teriparatide
Number analyzed (Participants) | 28
% change of Newtons | 17.43 (2.57)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, ANOVA

10. Secondary Outcome: Percent Change From Baseline in the Estimate of Bone Strength of Hip at Month 18 Endpoint
Description: Finite Element Analysis of computed tomography (CT) data from hip is used to estimate the strength of the proximal femur with a virtual sideways fall. Least squares (LS) mean of the percent change from baseline to 18 months is from an analysis of variance (ANOVA). The model included terms for investigator site and prior bisphosphonate use.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of Newtons
Arm/Group | Teriparatide
Number analyzed (Participants) | 25
% change of Newtons | 2.54 (1.18)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.045, ANOVA

11. Secondary Outcome: Percent Change From Baseline in Areal BMD at the Lumbar Spine at Month 18 and 24 Endpoint
Description: Areal BMD is a measure of the amount of mineral in a given area of bone. Least squares (LS) mean of the percent change from baseline to 18 and 24 months is from an analysis of variance (ANOVA). The model included terms for investigator site and prior bisphosphonate use.
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of g/square centimeter (g/cm²)
Arm/Group | Teriparatide
Number analyzed (Participants) | 29
% change of g/square centimeter (g/cm²)
  18 month percent change (n=28) | 7.215 (1.166)
  24 month percent change (n=25) | 8.702 (0.939)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for the percent change from baseline at 24 months

12. Secondary Outcome: Percent Change From Baseline in Areal BMD at the Femoral Neck at Month 18 and 24 Endpoint
Description: as for outcome 11
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of g/cm²
Arm/Group | Teriparatide
Number analyzed (Participants) | 29
% change of g/cm²
  18 month percent change (n=28) | 2.792 (0.998)
  24 month percent change (n=25) | 2.762 (1.312)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.011, ANOVA — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.049, ANOVA — P-value is for the percent change from baseline at 24 months

13. Secondary Outcome: Percent Change From Baseline in Areal BMD Responses at Total Hip at Month 18 and 24 Endpoint
Description: as for outcome 11
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of g/cm²
Arm/Group | Teriparatide
Number analyzed (Participants) | 29
% change of g/cm²
  18 month percent change (n=28) | 0.292 (0.747)
  24 month percent change (n=25) | 1.482 (0.836)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.700, ANOVA — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.092, ANOVA — P-value is for the percent change from baseline at 24 months

14. Secondary Outcome: Percent Change From Baseline in Areal BMD at ⅓ Distal Radius at Month 18 and 24 Endpoint
Description: as for outcome 11
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of g/cm²
Arm/Group | Teriparatide
Number analyzed (Participants) | 29
% change of g/cm²
  18 month percent change (n=28) | -2.068 (0.763)
  24 month percent change (n=25) | -2.733 (0.864)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.013, ANOVA — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.005, ANOVA — P-value is for the percent change from baseline at 24 months

15. Secondary Outcome: Percent Change From Baseline in Areal BMD at Ultra-Distal Radius at Month 18 and 24 Endpoint
Description: as for outcome 11
Time Frame: Baseline, 18, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of g/cm²
Arm/Group | Teriparatide
Number analyzed (Participants) | 29
% change of g/cm²
  18 month percent change (n=28) | -1.891 (1.122)
  24 month percent change (n=25) | 0.776 (0.975)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.106, ANOVA — P-value is for the percent change from baseline at 18 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.436, ANOVA — P-value is for the percent change from baseline at 24 months

16. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type I N-Terminal Propeptide (PINP) at Month 3, 6 and 24 Endpoint
Description: PINP is a measure of bone formation. Least squares (LS) mean of the percent change from baseline to 3, 6, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 3, 6, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of microgram/Liter (µg/L)
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of microgram/Liter (µg/L)
  3 month percent change (n=32) | 145.35 (23.36)
  6 month percent change (n=30) | 238.04 (44.29)
  24 month percent change (n=23) | 118.91 (22.72)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 3 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 6 months
Statistical Analysis 3: Comparison: Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 24 months

17. Secondary Outcome: Percent Change From Baseline in Serum Carboxyterminal Cross-Linking Telopeptide of Type I Collagen (CTX) at Month 3, 6 and 24 Endpoint
Description: CTX is a measure of bone resorption. Least squares (LS) mean of the percent change from baseline to 3, 6, 24 months is from a mixed model repeated measurements analysis. The model included terms for investigator site, prior bisphosphonate use, visit and baseline.
Time Frame: Baseline, 3, 6, 24 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: % change of nanogram/milliliter (ng/mL)
Arm/Group | Teriparatide
Number analyzed (Participants) | 32
% change of nanogram/milliliter (ng/mL)
  3 month percent change (n=32) | 63.53 (23.78)
  6 month percent change (n=30) | 102.56 (38.42)
  24 month percent change (n=23) | 48.28 (18.36)
Statistical Analysis 1: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.012, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 3 months
Statistical Analysis 2: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.012, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 6 months
Statistical Analysis 3: Comparison: Teriparatide; Test type: Superiority or Other; p = 0.016, Mixed Model Repeated Measurements — P-value is for the percent change from baseline at 24 months

ADVERSE EVENTS:
Arm/Group | Teriparatide
Serious Adverse Events (participants affected / at risk) | 5/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=35)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Injection site haematoma (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Weight decreased (Investigations) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (4)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days